CLINICAL TRIAL: NCT00535353
Title: A Phase I Study of AZD2281 in Combination With Irinotecan in Patients With Locally Advanced or Metastatic Incurable Colorectal Cancer
Brief Title: AZD2281 and Irinotecan in Treating Patients With Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I187; CAN-NCIC-IND187 (Registry Identifier: NCI US - Physician Data Query); IND187 (Other: NCIC CTG); CDR0000565189 (Other: PDQ)
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; stage III rectal cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: irinotecan hydrochloride — In Part A, a continuous oral AZD2281 dose will be given in combination with irinotecan given as a 90 minute infusion on day 1 every 21 days. In Part B, AZD2281 will be given on days 1-5 and irinotecan as a 90 minute infusion on day 3 each cycle. Cycles are repeated every 14 days.
Drug: olaparib — In Part A, a continuous oral AZD2281 dose will be given in combination with irinotecan given as a 90 minute infusion on day 1 every 21 days. In Part B, AZD2281 will be given on days 1-5 and irinotecan as a 90 minute infusion on day 3 each cycle. Cycles are repeated every 14 days.

SUMMARY:
RATIONALE: AZD2281 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AZD2281 together with irinotecan may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of AZD2281 and irinotecan in treating patients with locally advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the recommended phase II dose of AZD2281 and irinotecan hydrochloride in patients with locally advanced or metastatic colorectal cancer.
* To determine the safety, tolerability, toxicity profile, dose-limiting toxicities, and pharmacokinetic profile of this regimen.
* To assess the correlation, if any, between the toxicity profile and pharmacokinetics of this regimen.
* To assess, preliminarily, the antitumor activity of this regimen in patients with measurable disease.
* To demonstrate the pharmacodynamic activity of this regimen by establishing its effects in tumor biopsies, cheek swabs, and blood samples.
* To assess the correlation, if any, between patients with tumors demonstrating microsatellite instability and antitumor activity and pharmacodynamic effects of this regimen.
* To investigate the impact of common genetic polymorphisms of genes of relevant pathways (drug metabolism, DNA repair, and apoptosis) on outcome and toxicity as well as other pharmacodynamic effects.

OUTLINE: This is a multicenter, dose-escalation study of AZD2281 and irinotecan hydrochloride.

* Part I: Patients receive oral AZD2281 twice a day on days -7 to 21 in course 1 and on days 1-21 in all subsequent courses. Patients also receive irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 21 days (course 1 is 28 days) until the maximum tolerated dose is determined in the absence of disease progression or unacceptable toxicity.
* Part II: Patients then receive oral AZD2281 once daily on days 1-5 and irinotecan hydrochloride IV over 90 minutes on day 3 at the maximum tolerated dose determined in Part I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Patients undergo cheek swabs, tumor tissue, and blood sample collection periodically for pharmacokinetic, pharmacodynamic, and correlative studies.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer

  * Locally advanced and/or metastatic disease
  * Disease considered incurable
* Suitable for treatment with single agent irinotecan hydrochloride as a palliative intervention, as determined by the investigator
* Must have clinically and/or radiologically documented disease

  * Patients whose only evidence of disease progression is tumor marker elevation are not eligible
* Must have received no more than one prior oxaliplatin- and/or irinotecan hydrochloride-based chemotherapy regimen given either with adjuvant, neoadjuvant, or palliative intent

  * One additional adjuvant fluoropyrimidine (fluorouracil or capecitabine) regimen may have been given for relapsed or metastatic disease
* No untreated brain or meningeal metastases (CT scan required if there is a clinical suspicion of CNS disease)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2 times ULN (≤ 5 times ULN if liver metastasis is present)
* Serum creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after completion of study therapy
* Must reside within a 1½ hour drive from participating center
* No other invasive malignancies, unless curatively treated with no evidence of disease
* No GI tract disease resulting in an inability to absorb oral medication, including the following:

  * Uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
  * Post-surgical malabsorption characterized by uncontrolled diarrhea that results in weight loss and vitamin deficiency or requires IV hyperalimentation

    * Pancreatic enzyme supplementation is allowed
* No untreated and/or uncontrolled hypertension, cardiovascular conditions, and/or symptomatic cardiac dysfunction
* No active or uncontrolled infections
* No serious illnesses or medical conditions that would preclude study participation
* No known hypersensitivity to the study drugs or their components, atropine, or loperamide
* Not known to be homozygous for the UGT1A1*28 allele
* No known deficiency in glucuronidation of bilirubin, such as Gilbert's syndrome
* No neuropathy ≥ grade 2

  * Patients with persistent, stable, grade 3 sensory neuropathy, who meet other eligibility criteria may be allowed at the discretion of the investigator

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior PARP inhibitor
* No prior radical pelvic irradiation
* No prior radiotherapy to ≥ 25% of bone marrow stores
* Prior irinotecan hydrochloride allowed provided the drug was not discontinued due to toxic effects and the patient did not have severe irinotecan hydrochloride-related toxicity (grade 4 or requiring hospitalization)
* At least 21 days since prior radiotherapy (exceptions may be made for low-dose, nonmyelosuppressive radiotherapy)
* At least 30 days since prior chemotherapy
* At least 21 days since prior hormonal, immunologic, biologic, or signal transduction inhibitor therapies
* More than 3 weeks since prior and no other concurrent investigational drugs or anticancer therapy
* At least 14 days since prior major surgery

  * Wound healing must have occurred
* At least 14 days since prior and no concurrent CYP3A4 enzyme-inducing or -inhibiting drugs, including enzyme-inducing anticonvulsants, rifampin, rifabutin, St. John's wort, atazanavir, or ketoconazole

  * Dexamethasone is allowed for antiemetic prophylaxis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of AZD2281 and irinotecan hydrochloride | Nov 2011
  End of study
Safety | Nov 2011
  End of study
Tolerability | Nov 2011
  End of study
Dose-limiting toxicities | 2011-May-28
  Fatigue, Nausea, Dehydration and Anorexia.
Pharmacokinetic profile | Nov 2011
  End of study
Correlation, if any, between the toxicity profile and pharmacokinetics | Nov 2011
  End of study.

SECONDARY OUTCOMES:
Efficacy | Nov 2011
  End of study
Pharmacodynamic outcomes | Nov 2011
  End of study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric X. Chen, MD, PhD, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen EX, Jonker DJ, Siu LL, McKeever K, Keller D, Wells J, Hagerman L, Seymour L. A Phase I study of olaparib and irinotecan in patients with colorectal cancer: Canadian Cancer Trials Group IND 187. Invest New Drugs. 2016 Aug;34(4):450-7. doi: 10.1007/s10637-016-0351-x. Epub 2016 Apr 13. PMID 27075016